CLINICAL TRIAL: NCT00632320
Title: Effect of Continuous Positive Airway Pressure and Oxygen Concentration on Measurement of Rapid Shallow Breathing Index
Brief Title: Continuous Positive Airway Pressure and Oxygen Concentration on Measurement of Rapid Shallow Breathing Index
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Mauo-Ying Bien PhD, RPT, RRT/Assistant Professor, School of Respiratory Therapy, Taipei Medical University, Taipei, Taiwan
Other Study IDs: VGHIRB No.:93-09-02A; Grant 94CM-TMU-13; Grant NSC94-2314-B-038-039
Record Dates: First submitted 2008-03-02; First posted 2008-03-10 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-03

CONDITIONS: Acute Respiratory Failure
Keywords: Ventilator, mechanical; Ventilator weaning; Rapid shallow breathing index; Continuous positive airway pressure; Receiver operating characteristic curve; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- S, 1, A: group (success or failure), case number, measurement method

SUMMARY:
To compare the rapid shallow breathing index (RSBI) values, the incidence of adverse reactions, and the predictive accuracy measured under 5 different ventilator strategies in the same patient group.

DETAILED DESCRIPTION:
98 ready for weaning patients were included and divided into success (n=71) and failure (n=27) groups based upon their weaning outcome. Before weaning, the RSBI values were determined under the patients disconnecting from the ventilator (RA-no ventilator) and still connecting to the ventilator with 4 different settings (fraction of inspired oxygen (FiO2) 21 or 40% combined with continuous positive airway pressure (CPAP) 0 or 5 cm H2O). The patients were extubated after completing the weaning trials. Successful weaning was defined as patients free from the ventilator for over 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* intubated medical patients with mechanically ventilated more than 48 hours
* clinically ready for weaning
* Glasgow coma scales were at least 8
* their ventilator settings were: assist-controlled, pressure support (PS)or synchronized intermittent mandatory ventilation plus PS mode, FiO2 40% or less, positive end-expiratory pressure 5 cm H2O or less, and sensitivity setting on 1 L/min. Their arterial blood gases results were acceptable

Exclusion Criteria:

* having ongoing lung or neuromuscular disease and signs of increased intracranial pressure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: respiratory therapy intensive Care unit in a medical center
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2004-10; Primary Completion 2004-12 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The patients connecting or disconnecting to the ventilators affected the RSBI values but not their predictive accuracies. | Before the patient processing weaning trials

SECONDARY OUTCOMES:
Changes in FiO2 and CPAP settings have no effect on RSBI values but ventilator methods with FiO2 21% have higher incidence of adverse reactions. | Before the patient processing weaning trials

CONTACTS AND LOCATIONS:
Overall Officials: Mauo-Ying Bien, PhD, Principal Investigator — School of Respiratory Therapy, Taipei Medical University, Taipei, Taiwan, ROC
Locations (1):
- Respiratory Therapy Intensive Care Unit, Taipei Veterans General Hospital, Taipei, Taiwan